CLINICAL TRIAL: NCT06143683
Title: The Impact of Early Versus Late Upper Extremity Mobilization After Meshed / Sheet Split Thickness Skin Autograft on Wound Healing in Adult Burn Patients - A Single Center Non-Inferiority Randomized Clinical Trial
Brief Title: Early Versus Late Upper Extremity Mobilization After Meshed / Sheet Split Thickness Skin Autograft on Wound Healing in Adult Burn Patients
Acronym: EXTREMA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16820
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Burns
MeSH Terms: conditions — Burns | interventions — Early Ambulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Mobilization (Experimental)
  Interventions: Procedure: Early Mobilization
- Usual Care (Active Comparator)
  Interventions: Procedure: Late Mobilization

INTERVENTIONS:
Procedure: Early Mobilization — On post-operative day (POD) 1, active range of motion exercises of the elbow joint will be initiated under the observation and guidance of the physical therapy team. On POD 3, the patient will be transitioned to active as well as active-assisted range of motion exercises. The physical therapy team will provide an exercise sheet handout to patients (Appendix 5) and encourage patients to do the exercise for 10 repetitions, 2 times a day, holding each stretch for 30 seconds. On POD3, patients with non-meshed sheet hand grafts will undergo active range of motion exercises of the hands under the observation and guidance of the physical therapy team. On POD 5, the patient will be allowed to move the extremity as tolerated with no restrictions.
  Arms: Early Mobilization
Procedure: Late Mobilization — Following surgery, the patient's grafted upper extremity will be immobilized using an elbow flexion blocking splint. From POD 1 to 4, the patient's affected extremity will be kept elevated and immobilized with a flexion blocking splint. On POD 5, the patient will be allowed to move the extremity as tolerated with no restrictions. The physical therapy team will guide the patient on POD5 through range of motion exercises, starting with active, then active assisted, then passive as tolerated.
  Arms: Usual Care

SUMMARY:
STSGs are used to close wounds and minimize infections. After receiving a meshed or sheet split-thickness skin graft (STSG) to the upper extremity or hand for a thermal burn injury, burn surgeons use different methods to improve graft take and reduce complications. This includes different start dates and times for activity.

The goal of this clinical trial is to provide more evidence to improve rehabilitation procedures after STSG operations for patients with burn injuries. The main question[s] it aims to answer are:

* To determine if early mobilization is non-inferior to late mobilization of the upper extremity after meshed STSG with regards to wound healing in adult burn patients.
* To determine if early mobilization is non-inferior to late mobilization of the upper extremity after sheet STSG with regards to wound healing in adult burn patients

Participants will be assigned randomly (like flipping a coin) to one of two groups: early mobilization and late mobilization. Mobilization is the range of motion exercises performed under the supervision of the physical therapy team. Researchers will compare early and late mobilization to see if there are differences in wound healing, range of motion, local and systemic complications, and discharge outcomes.

Participants will be asked to:

* Early mobilization group: begin mobilization of their upper extremity one day after their STSG operation. If their burn includes a graft to your hand, early mobilization of this area will begin three days after their STSG operation.
* Late mobilization group: elevate their elbow in a splint to limit movement until five days after their operation and begin mobilization five days after their STSG operation.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years and older at the time of surgery.
* Injury: Acute (within 72h of injury) thermal flame or scald burn.
* Surgery: Skin split-thickness meshed autograft (STSG) and/or sheet split thickness autograft (STSG) applied directly on the wound bed.
* Location:

  1. Upper extremity burn - distal to the axilla and proximal to the wrist. The axilla is a difficult area to graft due to its three-dimensional configuration, hence the healing of this area is not comparable to others.
  2. The hand that will undergo sheet STSG

Exclusion Criteria:

* Injury: Electrical and chemical burn. The pathophysiology of electrical or chemical burns is not comparable to flame or scald burns, hence their exclusion.
* Location: Autograft exclusively to the wrist, axilla, or non-upper extremity. The wrist is a sensitive areas with many joints in close proximity. The loss of graft in this area can be devastating to the patient and will therefore be evaluated only once we have evidence to support the safety of mobilization in upper extremity grafts.
* Patients on vasopressors the day of the operation. Vasopressors cause peripheral vasoconstriction, leading to decreased wound healing capacity. Patients on vasopressors are also usually systemically unwell and should therefore not be included in an elective clinical trial on extremity mobilization.
* Pre-existing comorbidities causing upper extremity mobility restrictions.
* Patient unable to comply with mobilization protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Wound healing measured as percent graft take on POD5 (± 2 days) | From autografting until five days afterwards

SECONDARY OUTCOMES:
Percent graft healed at POD 14 (± 2 days) | From autografting until 14 days afterwards
  Photographs used to evaluate the primary and secondary wound healing outcomes will be reviewed by a blinded and trained researcher to estimate the percentage of the grafted area that has healed. The photographs will be taken by a trained member of the Hamilton General Hospital Burn Unit if the patient is admitted, and by a trained member of the burn clinic if the patient is discharged and presenting for follow-up.
Incidence of post-operative local complications (seroma, hematoma, infection, graft loss) or systemic complications (infection, deep vein thrombosis, pulmonary embolism, mortality) | From autografting until 14 days afterwards
Severity of graft site pain | From autografting until five days afterwards
  Patients will self-report graft site pain at rest and with mobilization using the Visual Analogue Pain Scale. The scale is scored from 0 (no pain) to 10 (worst possible pain).
Range of motion of the elbow joint | From autografting until 14 days afterwards
  Active range of motion (ROM) for flexion and extension of the elbow will be measured using a goniometer.
Range of motion of the hand | From autografting until 14 days afterwards
  Active range of motion (ROM) for flexion and extension of the hand joints (metacarpals, IP, PIP, and DIP joints) will be measured using a goniometer.
Days to discharge from the Burn Unit | From admission to the burn unit until discharge (approximately 2 days for every 1% total body surface area burn).
  The staff physician responsible for the care of the patient in collaboration with the members of the multidisciplinary team will evaluate on a daily basis the patient readiness for discharge based on a list of criteria and determine most appropriate discharge location.
Days between admission to the burn unit and the date of discharge. | From admission to the burn unit until discharge (approximately 2 days for every 1% total body surface area burn).

CONTACTS AND LOCATIONS:
Overall Officials: Shahriar Shahrokhi, MD, Principal Investigator — Hamilton Health Sciences Corporation